CLINICAL TRIAL: NCT02624648
Title: Effects of Lepidium Meyenii Walp (Peruvian Maca) on Sexual Function in Postmenopausal
Brief Title: Effects of Lepidium Meyenii Walp on Sexual Function in Postmenopausal Women
Acronym: maca
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Vale do Sapucai (Other)
Collaborators: Irmandade da Santa Casa de Misericordia de Sao Paulo (Other)
Responsible Party: Principal Investigator, Benedito Fabiano dos Reis, MD, Universidade do Vale do Sapucai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAAE 43373915.3.0000.5479
Record Dates: First submitted 2015-11-30; First posted 2015-12-08 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Sexual Dysfunction, Physiological
Keywords: Sexual Dysfunction; Postmenopausal women; Sexual desire
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — MacA protein, E coli

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Group (Placebo Comparator): The effects of Placebo on sexual function, desire and depression in postmenopausal women.
  The Female Sexual Function Index (FSFI) and the Female Intervention Efficacy Index Questionnaire (FIEI).
  The Beck Depression Inventory II will be used to ward off depression
  Interventions: Behavioral: The Female Sexual Function Index (FSFI); Behavioral: The Female Intervention Efficacy Index (FIEI); Behavioral: The Beck Depression Inventory II; Drug: Placebo
- Maca (Lepidium Meyenii Walp) Group (Experimental): The effects of Lepidium Meyenii Walp on sexual function, desire and depression in postmenopausal women.
  The Female Sexual Function Index (FSFI) and the Female Intervention Efficacy Index Questionnaire (FIEI).
  The Beck Depression Inventory II will be used to ward off depression
  Interventions: Behavioral: The Female Sexual Function Index (FSFI); Behavioral: The Female Intervention Efficacy Index (FIEI); Behavioral: The Beck Depression Inventory II; Drug: Lepidium Meyenii Walp

INTERVENTIONS:
Behavioral: The Female Sexual Function Index (FSFI) — The Female Sexual Function Index (FSFI) Questionnaire to evaluate the sexual function
Behavioral: The Female Intervention Efficacy Index (FIEI) — The Female Intervention Efficacy Index Questionnaire (FIEI) to evaluate the sexual function
Behavioral: The Beck Depression Inventory II — The Beck Depression Inventory II will be used to evaluate or ward off depression
Drug: Lepidium Meyenii Walp — They will receive a capsule of Lepidium Meyenii Walp twice a day for 120 days
  Other Names: Maca
  Arms: Maca (Lepidium Meyenii Walp) Group
Drug: Placebo — They will receive a capsule of Placebo twice a day for 120 days
  Arms: Placebo Group

SUMMARY:
Objective: To study the effects of Lepidium Meyenii in sexual function of postmenopausal women.

Method: It will be held a clinical, prospective, randomized, double-blind, placebo-controlled study with 144 postmenopausal women with sexual dysfunction, treated at Menopause Clinic at the Faculty of Medical Sciences of Santa Casa de São Paulo and in the Vale do Sapucai University. All women sign the Consent Form Term. The study will be conducted in accordance with the protocol and principles of the Declaration Helsinki (Version 1996), according to International Conference on Harmonization and Tripartite Guidelines for good clinical practice and regulatory requirements. The protocol was approved by the Ethics Committee of the Faculty of Medical Sciences of Santa Casa de São Paulo.

Hypothesis: It is expected to be an improvement of sexual function in postmenopausal women.

DETAILED DESCRIPTION:
It will be a prospective, randomized, double-blind, placebo-controlled study with 144 postmenopausal women with sexual dysfunction, met in Menopause Clinic at the Faculty of Medical Sciences of Santa Casa de São Paulo and in the Vale do Sapucai University. All women signed the Informed Consent. The study will be conducted in accordance with the protocol and principles set out in Declaration of Helsinki (1996 version), according to International Conference on Harmonization and Tripartite Guidelines for good practice clinics and applicable regulatory requirements.

The protocol was submitted and approved by the Ethics Committee, Faculty of Medical Sciences Committee Santa Casa de São Paulo. The diagnosis of sexual dysfunction will be done by a sexologist physician experienced and trained in the diagnosis of female sexual disorders through a structured clinical interview, a list of sexual symptoms. It will be oriented to avoid further consumption of diet or another type of herbal medicine during the study. After the interview, signing the Informed Consent and they will be informed about the randomization. Interview with sexological questionnaires will be applied used in Sexology Clinic, Faculty of Medical Sciences of Santa Casa de São Paulo and Vale do Sapucai University, with the purpose of obtaining data sociodemographic. The Female Sexual function Index (FSFI) and the Female Intervention Efficacy Index questionnaire (FIEI). When necessary, the Beck Depression Inventory II (Cunha 2001) will be used to ward off depression, which will be applied by enabled professional. The application will be individually and by the same researcher. The results will be analyzed and interpreted in the light of the theoretical framework of socio-historical psychology, this theory of knowledge, is associated with the understanding of the culture of the structure, social organization and the rescue human subjectivity.

ELIGIBILITY:
Inclusion Criteria:

* The postmenopausal women with full autonomy, with one year or more of amenorrhea and follicle stimulating hormone (FSH) > 30 milli-International unit/mL
* Women who are not regularly practicing sexual activity will be included because the desire domain is subject to the same evaluation in this situation
* Estrogen and progesterone were permitted if the dose had been stable for six months prior to screening

Exclusion Criteria:

* Cardiac, renal and hepatic diseases
* Diabetes mellitus
* Cognitive disorders
* Hormone-dependent tumor
* History of psychiatric illness current and/or past, regular use of two or more doses of alcohol by day (dose = 12 grams of pure alcohol, which corresponds to 330 mL of beer, 100 mL wine, 30 mL of distilled World Health Organization standard dose) leading to impairment or clinically significant distress (DSM-5)
* Consumption of Maca supplements or any other nutritional supplement known to cause changes in sexual function
* Use of any drug that, in the opinion of the investigator, may affect sexual function or any of the following medications: anti-epileptics, cytochrome P450 isoform 3A4 (CYP3A4) inducers
* Dopamine agonists and other parkinsonian drugs
* Metoclopramide
* Androgens and antiandrogens, the anti-oestrogens
* Fluoxetine or any hormonal implant long-acting in 30 days before the exam
* Analogues of gonadotropin-releasing hormone and other hormones and inhibitors
* Benzodiazepines prescribed for insomnia
* Sedatives and hypnotics
* Antidepressants
* Antipsychotics, mood stabilizers, narcotics (except when used to relieve short-term pain),
* Lubricants/moisturizers that contain substances that promote heating and/or vaginal stimulators

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
FSFI Questionnaire to evaluate the sexual function | 120 days
  To study the effects of Lepidium meyenii and placebo on sexual function in postmenopausal women

SECONDARY OUTCOMES:
FIEI Questionnaire to evaluate the sexual desire | 120 days
  To study the effects of Lepidium meyenii and placebo on sexual desire in postmenopausal women

OTHER OUTCOMES:
The Beck Depression Inventory II to evaluate depression | 120 days
  It will be used to evaluate or ward off depression

CONTACTS AND LOCATIONS:
Overall Officials: Fabiola SM Campos, MD, Study Director — Universidade do Vale do Sapucai; Sonia Maria R Rosa Lima, PhD, Principal Investigator — Santa Casa of São Paulo
Locations (1):
- Vale Do Sapucai University (Univas), Pouso Alegre, Minas Gerais, Brazil

REFERENCES:
- [Result] Dailey RK, Neale AV, Northrup J, West P, Schwartz KL. Herbal product use and menopause symptom relief in primary care patients: a MetroNet study. J Womens Health (Larchmt). 2003 Sep;12(7):633-41. doi: 10.1089/154099903322404285. PMID 14583104
- [Result] Geller SE, Studee L. Botanical and dietary supplements for menopausal symptoms: what works, what does not. J Womens Health (Larchmt). 2005 Sep;14(7):634-49. doi: 10.1089/jwh.2005.14.634. PMID 16181020
- [Result] Kronenberg F, Fugh-Berman A. Complementary and alternative medicine for menopausal symptoms: a review of randomized, controlled trials. Ann Intern Med. 2002 Nov 19;137(10):805-13. doi: 10.7326/0003-4819-137-10-200211190-00009. PMID 12435217
- [Result] van der Sluijs CP, Bensoussan A, Liyanage L, Shah S. Women's health during mid-life survey: the use of complementary and alternative medicine by symptomatic women transitioning through menopause in Sydney. Menopause. 2007 May-Jun;14(3 Pt 1):397-403. doi: 10.1097/01.gme.0000236937.36078.f4. PMID 17202872
- [Result] Minelli C, Abrams KR, Sutton AJ, Cooper NJ. Benefits and harms associated with hormone replacement therapy: clinical decision analysis. BMJ. 2004 Feb 14;328(7436):371. doi: 10.1136/bmj.328.7436.371. PMID 14962874
- [Result] Low Dog T. Menopause: a review of botanical dietary supplements. Am J Med. 2005 Dec 19;118 Suppl 12B:98-108. doi: 10.1016/j.amjmed.2005.09.044. PMID 16414334
- [Result] Chung F, Rubio J, Gonzales C, Gasco M, Gonzales GF. Dose-response effects of Lepidium meyenii (Maca) aqueous extract on testicular function and weight of different organs in adult rats. J Ethnopharmacol. 2005 Apr 8;98(1-2):143-7. doi: 10.1016/j.jep.2005.01.028. PMID 15763375
- [Result] Meissner HO, Kapczynski W, Mscisz A, Lutomski J. Use of gelatinized maca (lepidium peruvianum) in early postmenopausal women. Int J Biomed Sci. 2005 Jun;1(1):33-45. PMID 23674952
- [Result] Gonzales GF, Cordova A, Gonzales C, Chung A, Vega K, Villena A. Lepidium meyenii (Maca) improved semen parameters in adult men. Asian J Androl. 2001 Dec;3(4):301-3. PMID 11753476
- [Result] Gonzales GF, Ruiz A, Gonzales C, Villegas L, Cordova A. Effect of Lepidium meyenii (maca) roots on spermatogenesis of male rats. Asian J Androl. 2001 Sep;3(3):231-3. PMID 11561196
- [Result] Gonzales GF, Cordova A, Vega K, Chung A, Villena A, Gonez C, Castillo S. Effect of Lepidium meyenii (MACA) on sexual desire and its absent relationship with serum testosterone levels in adult healthy men. Andrologia. 2002 Dec;34(6):367-72. doi: 10.1046/j.1439-0272.2002.00519.x. PMID 12472620
- [Result] Gonzales GF, Cordova A, Vega K, Chung A, Villena A, Gonez C. Effect of Lepidium meyenii (Maca), a root with aphrodisiac and fertility-enhancing properties, on serum reproductive hormone levels in adult healthy men. J Endocrinol. 2003 Jan;176(1):163-8. doi: 10.1677/joe.0.1760163. PMID 12525260
- [Result] Gonzales GF, Gasco M, Cordova A, Chung A, Rubio J, Villegas L. Effect of Lepidium meyenii (Maca) on spermatogenesis in male rats acutely exposed to high altitude (4340 m). J Endocrinol. 2004 Jan;180(1):87-95. doi: 10.1677/joe.0.1800087. PMID 14709147
- [Result] Gonzales GF, Miranda S, Nieto J, Fernandez G, Yucra S, Rubio J, Yi P, Gasco M. Red maca (Lepidium meyenii) reduced prostate size in rats. Reprod Biol Endocrinol. 2005 Jan 20;3:5. doi: 10.1186/1477-7827-3-5. PMID 15661081
- [Result] Oshima M, Gu Y, Tsukada S. Effects of Lepidium meyenii Walp and Jatropha macrantha on blood levels of estradiol-17 beta, progesterone, testosterone and the rate of embryo implantation in mice. J Vet Med Sci. 2003 Oct;65(10):1145-6. doi: 10.1292/jvms.65.1145. PMID 14600359
- [Result] Zheng BL, He K, Kim CH, Rogers L, Shao Y, Huang ZY, Lu Y, Yan SJ, Qien LC, Zheng QY. Effect of a lipidic extract from lepidium meyenii on sexual behavior in mice and rats. Urology. 2000 Apr;55(4):598-602. doi: 10.1016/s0090-4295(99)00549-x. PMID 10736519
- [Result] Cicero AF, Bandieri E, Arletti R. Lepidium meyenii Walp. improves sexual behaviour in male rats independently from its action on spontaneous locomotor activity. J Ethnopharmacol. 2001 May;75(2-3):225-9. doi: 10.1016/s0378-8741(01)00195-7. PMID 11297856
- [Result] Ruiz-Luna AC, Salazar S, Aspajo NJ, Rubio J, Gasco M, Gonzales GF. Lepidium meyenii (Maca) increases litter size in normal adult female mice. Reprod Biol Endocrinol. 2005 May 3;3:16. doi: 10.1186/1477-7827-3-16. PMID 15869705
- [Result] Valentova K, Buckiova D, Kren V, Peknicova J, Ulrichova J, Simanek V. The in vitro biological activity of Lepidium meyenii extracts. Cell Biol Toxicol. 2006 Mar;22(2):91-9. doi: 10.1007/s10565-006-0033-0. Epub 2006 Mar 9. PMID 16528448
- [Result] Bogani P, Simonini F, Iriti M, Rossoni M, Faoro F, Poletti A, Visioli F. Lepidium meyenii (Maca) does not exert direct androgenic activities. J Ethnopharmacol. 2006 Apr 6;104(3):415-7. doi: 10.1016/j.jep.2005.09.028. Epub 2005 Oct 18. PMID 16239088
- [Result] Freeman EW, Sammel MD, Liu L, Gracia CR, Nelson DB, Hollander L. Hormones and menopausal status as predictors of depression in women in transition to menopause. Arch Gen Psychiatry. 2004 Jan;61(1):62-70. doi: 10.1001/archpsyc.61.1.62. PMID 14706945
- [Result] Rubio J, Caldas M, Davila S, Gasco M, Gonzales GF. Effect of three different cultivars of Lepidium meyenii (Maca) on learning and depression in ovariectomized mice. BMC Complement Altern Med. 2006 Jun 23;6:23. doi: 10.1186/1472-6882-6-23. PMID 16796734
- [Result] Bosworth HB, Bastian LA, Kuchibhatla MN, Steffens DC, McBride CM, Skinner CS, Rimer BK, Siegler IC. Depressive symptoms, menopausal status, and climacteric symptoms in women at midlife. Psychosom Med. 2001 Jul-Aug;63(4):603-8. doi: 10.1097/00006842-200107000-00013. PMID 11485114
- [Result] Dennerstein L, Alexander JL, Kotz K. The menopause and sexual functioning: a review of the population-based studies. Annu Rev Sex Res. 2003;14:64-82. PMID 15287158
- [Result] Gonzales GF, Gonzales C, Gonzales-Castaneda C. Lepidium meyenii (Maca): a plant from the highlands of Peru--from tradition to science. Forsch Komplementmed. 2009 Dec;16(6):373-80. doi: 10.1159/000264618. Epub 2009 Dec 16. PMID 20090350
- [Result] Berman LA, Berman JR, Werbin T, Chabra S, Goldstein I. The use of the Female Intervention Efficacy Index (FIEI) as an immediate outcome measure of medical intervention to treat female sexual dysfunction. J Sex Marital Ther. 2001 Oct-Dec;27(5):427-33. doi: 10.1080/713846821. PMID 11554203